CLINICAL TRIAL: NCT01824303
Title: A Phase 2 Multicenter, Randomized, Double-Blinded, Placebo-Controlled Study Evaluating Safety, Tolerability and Efficacy of LiRIS® 400 mg in Women With Interstitial Cystitis Followed by an Open Label Extension
Brief Title: Safety, Tolerability and Efficacy Study of LiRIS® 400 mg in Women With Interstitial Cystitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was terminated early due to company decision.
Sponsor: Allergan (Industry)
Collaborators: TARIS Biomedical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TAR-100-202
Record Dates: First submitted 2013-03-31; First posted 2013-04-04 (Estimated); Results first posted 2015-11-26 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2015-12

CONDITIONS: Interstitial Cystitis
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LiRIS 400 mg (Experimental): LiRIS 400 mg: investigational drug-delivery system which contains Lidocaine; the system remains in the bladder for 14 days. If eligible, participants could participate in the Open Label Extension where all participants were treated with LiRIS 400 mg.
  Interventions: Drug: LiRIS 400 mg
- LiRIS Placebo (Placebo Comparator): LiRIS Placebo: investigational drug-delivery system which contains Lactose and no Lidocaine; the system remains in the bladder for 14 days. If eligible, participants could participate in the Open Label Extension where all participants were treated with LiRIS 400 mg.
  Interventions: Other: LiRIS Placebo

INTERVENTIONS:
Drug: LiRIS 400 mg — LiRIS 400 mg contains lidocaine which is gradually released into the bladder over 14 days.
  Arms: LiRIS 400 mg
Other: LiRIS Placebo — LiRIS Placebo contains lactose, inactive substance.
  Arms: LiRIS Placebo

SUMMARY:
The purposes of the study is to determine if LiRIS®, an investigational drug-delivery system, is safe and tolerable in women with Interstitial Cystitis (IC), and to evaluate any change in IC symptoms following LiRIS administration.

DETAILED DESCRIPTION:
The study is conducted in 2 parts: a randomized, blinded part in which subjects are assigned randomly (by chance) to LiRIS 400 mg or LiRIS placebo; subjects who complete this part and are eligible to continue, may participate in the open-label part in which all subjects receive LiRIS 400 mg.

In both parts of the study (blinded and open-label), LiRIS is inserted into the bladder during cystoscopy, remains in the bladder for 14 days, and is removed during cystoscopy. In addition to the 14 day period with the LiRIS/LiRIS Placebo, there is a screening period of up to 2 weeks and a follow up period of 4 weeks.

ELIGIBILITY:
Inclusion Criteria

Blinded study:

* Women age 18 and over
* Diagnosed with Interstitial Cystitis as defined by protocol
* Able to report IC symptoms of bladder pain, voiding habits, as required by protocol, and record in diary
* Able to comply with visit schedule and diary completion at home

Open-label Extension:

* Must have completed the blinded study prior to screening for the Open-label extension

Exclusion Criteria (Blinded and Open-Label Extension):

* Pregnant or lactating women
* History or presence of any condition that would make it difficult to accurately evaluate bladder symptoms
* Bladder or urethral abnormality that would prevent safe insertion of investigational product
* Requiring medication not allowed per study protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-03; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Curtis Nickel, MD, Principal Investigator — Queen's University/Kingston General Hospital/Ontario Canada
Locations (17):
- United States (15):
  - Citrus Valley Medical Research , Inc., Glendora, California
  - Atlantic Urological Associates, Daytona Beach, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - The UrogynecologyCenter, LLC, Overland Park, Kansas
  - Female Pelvic Medicine & Urogynecology Institute of MI, Grand Rapids, Michigan
  - William Beaumont Hospitals, Royal Oak, Michigan
  - North Shore - Long Island Jewish Heath System - Monter Cancer Center, New Hyde Park, New York
  - Premier Medical Group of the Hudson Valley PC, Newburgh, New York
  - Premier Medical Group of the Hudson Valley PC, Poughkeepsie, New York
  - Alliance Urology Specialists, PA, Greensboro, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - MetroHealth Medical Center, Cleveland, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Volunteer Research Group, University of Tennessee Medical Center, Knoxville, Tennessee
- Canada (2):
  - Exdeo Clinical Research Inc., Abbotsford, British Columbia
  - Centre for Applied Urological Research, Kingston, Ontario

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 31 participants signed the informed consent form and were enrolled in the study, 30 participants had the investigational product inserted and are included the Intent-to-treat Population.
Groups:
- LiRIS 400 mg: LiRIS 400 mg: investigational drug-delivery system which contains Lidocaine; the system remains in the bladder for 14 days.
- LiRIS Placebo: LiRIS Placebo: investigational drug-delivery system which contains Lactose and no Lidocaine; the system remains in the bladder for 14 days.
Period: Randomized Study
Arm/Group | LiRIS 400 mg | LiRIS Placebo
Started | 16 | 14
Completed | 14 | 13
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Other Miscellaneous Reasons | 1 | 0
Period: Open Label Extension
Arm/Group | LiRIS 400 mg | LiRIS Placebo
Started | 12 (2 participants completed the Randomized Study but did not enter the Open Label Extension.) | 11 (2 participants completed the Randomized Study but did not enter the Open Label Extension.)
Completed | 12 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LiRIS 400 mg | LiRIS Placebo | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.7 (14.13) | 42.1 (10.54) | 41.9 (12.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 30
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Participant Reported Average Bladder Pain on a Numerical Rating Scale (NRS)
Description: Participants rated their bladder pain over the previous 24 hours in an electronic diary using a horizontal line NRS by putting a mark on the line where: 0 (the far left of the line)=no pain to 10 (far right of the line)=worst pain imaginable. Bladder pain was averaged over a period of 3 days. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Day 12
Population: Intent-to-treat (ITT) population included all randomized participants.
Measure: Mean (Standard Deviation); unit: unit on a scale
Arm/Group | LiRIS 400 mg | LiRIS Placebo
Number analyzed (Participants) | 16 | 14
unit on a scale
  Baseline | 7.04 (0.750) | 7.67 (1.067)
  Change from Baseline at Day 12 | -1.44 (1.584) | -2.50 (2.723)

2. Secondary Outcome: Change From Baseline in Total Daily Voids
Description: Participants recorded number of daily voids (day-time and night-time daily voids) in a 3 day Voiding Frequency electronic diary. The total number of daily voids was averaged over a period of 3 full days. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Day 27
Population: Participants from the ITT population, all randomized participants, with data available for analyses.
Measure: Mean (Standard Deviation); unit: voids
Arm/Group | LiRIS 400 mg | LiRIS Placebo
Number analyzed (Participants) | 16 | 14
voids
  Baseline | 13.4 (6.52) | 14.9 (7.81)
  Change from Baseline at Day 27 (n=15,14) | -2.9 (4.64) | -3.3 (4.93)

3. Secondary Outcome: Change From Baseline in Night-Time Daily Voids
Description: Participants recorded number of night-time daily voids in a 3 day Voiding Frequency electronic diary. The total number of night-time daily voids was averaged over a period of 3 days. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Day 27
Population: Participants from the ITT population, all randomized participants, with data available for analyses.
Measure: Mean (Standard Deviation); unit: voids
Arm/Group | LiRIS 400 mg | LiRIS Placebo
Number analyzed (Participants) | 16 | 14
voids
  Baseline | 2.4 (2.56) | 2.1 (2.37)
  Change from Baseline at Day 27 (n=15,14) | -0.5 (2.09) | -0.9 (2.00)

4. Secondary Outcome: Change From Baseline in Average Void Volume Per Micturition
Description: Participants recorded the amount of each void in millimeters (mL) in an electronic diary. The total amount of void per micturition (each void) was averaged over a period of 24 days. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Day 27
Population: Participants from the ITT population, all randomized participants, with data available for analyses.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | LiRIS 400 mg | LiRIS Placebo
Number analyzed (Participants) | 16 | 14
mL
  Baseline | 141.1 (80.26) | 120.3 (73.06)
  Change from Baseline at Day 27 (n=14,12) | -2.2 (73.31) | -0.5 (43.86)

5. Secondary Outcome: Change From Baseline in Post-Void Bladder Pain
Description: Participants rated their bladder pain immediately completing voiding in an electronic diary using a horizontal line NRS by putting a mark on the line where: 0 (the far left of the line)=no pain to 10 (far right of the line)=worst pain imaginable. The average of the data from the first 5 voids prior to Baseline and the 3 days prior to Day 12 were averaged for analyses. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Day 27
Population: Participants from the ITT population, all randomized participants, with data available for analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LiRIS 400 mg | LiRIS Placebo
Number analyzed (Participants) | 16 | 14
units on a scale
  Baseline (n=13,11) | 4.86 (1.857) | 6.17 (1.925)
  Change from Baseline at Day 27 (n=12,10) | -1.05 (1.805) | -1.69 (1.997)

6. Secondary Outcome: Change From Baseline in O'Leary-Sant Interstitial Cystitis Symptom Index (ICSI) Score
Description: The ICSI is a participant reported questionnaire to rate their symptoms by answering 4 questions. Question (Q) 1 and 2 (urine urgency) using a 6-point scale where: 0=Not at All to 5=Almost Always. Q3 (night-time voids) using a 6-point scale where: 0=None to 5=5 or More Times. Q4 (pain and burning) using a 6-point scale where: 0=Not at All to 5=Usually. The total score is the sum of the individual scores for a total possible score of 0 (best) to 20 (worst). A negative change from Baseline indicates improvement.
Time Frame: Baseline, Day 27
Population: Participants from the ITT population, all randomized participants, with data available for analyses.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LiRIS 400 mg | LiRIS Placebo
Number analyzed (Participants) | 16 | 14
score on a scale
  Baseline | 14.1 (3.70) | 14.2 (2.73)
  Change from Baseline at Day 27 (n=14,12) | -1.4 (3.79) | -2.8 (3.04)

7. Secondary Outcome: Change From Baseline in O'Leary-Sant Interstitial Cystitis Problem Index (ICPI) Score
Description: The ICPI is a participant reported questionnaire to rate their problems in the following 4 areas: Frequent urination; Getting up at Night to Urinate: Urination with little warning; Burning pain and discomfort. Questions are answered on a 5-point scale where: 0=No Problem to 4=Big Problem. The total score is the sum of the individual scores for a total possible score of 0 (best) to 20 (worst). A negative change from Baseline indicates improvement.
Time Frame: Baseline, Day 27
Population: Participants from the ITT population, all randomized participants, with data available for analyses.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LiRIS 400 mg | LiRIS Placebo
Number analyzed (Participants) | 16 | 14
score on a scale
  Baseline | 12.4 (2.87) | 13.9 (1.66)
  Change from Baseline at Day 27 (n=14,12) | -1.3 (3.52) | -3.2 (3.46)

8. Secondary Outcome: Change From Baseline in Bladder Pain/Interstitial Cystitis Symptom Score (BPIC-SS)
Description: The BPIC-SS is a participant reported questionnaire consisting of 8 items. Questions (Q) 1-5 (How often urination because of pain; Need to urinate after just urinating; How often urination to avoid worse pain; How often feeling of pressure in bladder; How often pain in bladder) answered on a 5-point scale where: 0=Never to 4=Always. Q 6-7 (Bothered by frequent Day-time urination; Bothered by Night-time urination) answered on a 5-point scale where: 0=Not At All to 4=A Great Deal. Q8 (pain) rated on a NRS by putting a mark on the line where: 0 (the far left of the line)=no pain to 10 (far right of the line)=worst pain imaginable. The Total Score is the sum of the individual questionnaire of all 8 items for a total possible score of 0 (best) to 38 (worst). A negative change indicates improvement.
Time Frame: Baseline, Day 27
Population: Participants from the ITT population, all randomized participants, with data available for analyses.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LiRIS 400 mg | LiRIS Placebo
Number analyzed (Participants) | 16 | 14
score on a scale
  Baseline (n=16,13) | 28.8 (4.16) | 31.2 (3.00)
  Change from Baseline at Day 27 (n=14,12) | -4.0 (5.75) | -7.1 (7.81)

9. Secondary Outcome: Change From Baseline in Brief Pain Inventory (BPI)
Description: The BPI is a 7-item participant completed questionnaire. The participant answered questions as to how pain interfered with: General Activity, Mood, Walking Ability, Normal work, Relations with other people, Sleep and Enjoyment of life. Questions were answered on an 11-point scale where: 0=Does not interfere to 10=Completely interferes. The total score is the average of the individual questionnaire items for a total possible score of 0 (best) to 10 (worst). A negative change from Baseline indicates improvement.
Time Frame: Baseline, Day 27
Population: Participants from the ITT population, all randomized participants, with data available for analyses.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LiRIS 400 mg | LiRIS Placebo
Number analyzed (Participants) | 16 | 14
score on a scale
  Baseline (n=16,13) | 6.5 (1.10) | 7.2 (1.99)
  Change from Baseline at Day 27 (n=14,12) | -1.2 (2.52) | -2.3 (2.21)

ADVERSE EVENTS:
Groups:
- LiRIS 400 mg_Randomized Study: LiRIS 400 mg: investigational drug-delivery system which contains Lidocaine; the system remains in the bladder for 14 days in the randomized study.
- LiRIS Placebo_Randomized Study: LiRIS Placebo: investigational drug-delivery system which contains Lactose and no Lidocaine; the system remains in the bladder for 14 days in the randomized study.
- LiRIS 400 mg_Open Label Extension: LiRIS 400 mg: investigational drug-delivery system which contains Lidocaine; the system remains in the bladder for 14 days in the randomized study then LiRIS 400 mg in the Open Label Extension.
- LiRIS Placebo/LiRIS 400 mg _Open Label Extension: LiRIS Placebo: investigational drug-delivery system which contains Lactose and no Lidocaine; the system remains in the bladder for 14 days in the randomized study then LiRIS 400 mg in the Open Label Extension.
Arm/Group | LiRIS 400 mg_Randomized Study | LiRIS Placebo_Randomized Study | LiRIS 400 mg_Open Label Extension | LiRIS Placebo/LiRIS 400 mg _Open Label Extension
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14 | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 11/16 | 12/14 | 6/12 | 6/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LiRIS 400 mg_Randomized Study (N=16) | LiRIS Placebo_Randomized Study (N=14) | LiRIS 400 mg_Open Label Extension (N=12) | LiRIS Placebo/LiRIS 400 mg _Open Label Extension (N=11)
Dysuria (Renal and urinary disorders) | 4 | 4 | 0 | 2
Bladder pain (Renal and urinary disorders) | 2 | 3 | 0 | 1
Bladder discomfort (Renal and urinary disorders) | 2 | 2 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 2 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 2 | 0 | 0
Urethral pain (Renal and urinary disorders) | 2 | 0 | 1 | 1
Bladder spasm (Renal and urinary disorders) | 0 | 1 | 0 | 0
Cystitis interstitial (Renal and urinary disorders) | 1 | 0 | 1 | 2
Micturition urgency (Renal and urinary disorders) | 1 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 2 | 2 | 1
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0
Genital herpes (Infections and infestations) | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 2
Tooth abscess (Infections and infestations) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 0
Pallor (Vascular disorders) | 0 | 1 | 0 | 0
Allergy to arthropod bite (Immune system disorders) | 0 | 1 | 0 | 0
Allergy to arthropod sting (Immune system disorders) | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 0
Residual urine volume increased (Investigations) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 1
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Pelvic discomfort (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 1 | 0
Urethritis noninfective (Renal and urinary disorders) | 0 | 0 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vitamin D decreased (Investigations) | 0 | 0 | 0 | 1
Burning sensation (Nervous system disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Due to technical issues with the patient electronic diary used for the collection of the outcome measures data, as well as the small evaluable sample size and large variability, the efficacy data should be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.